CLINICAL TRIAL: NCT02016729
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AMG 232 Alone and in Combination With Trametinib in Adult Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Phase 1b Study Evaluating AMG 232 Alone and in Combination With Trametinib in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120234
Record Dates: First submitted 2013-11-21; First posted 2013-12-20 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Advanced Malignancy; Cancer; Oncology; Oncology Patients; Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Neoplasms; Leukemia, Myeloid, Acute | interventions — 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 232 (Experimental): AMG 232 is an anti-cancer agent
  Interventions: Drug: AMG 232; Drug: Trametinib
- AMG 232 & Trametinib (Experimental): AMG 232 and Trametinib are anti cancer agents
  Interventions: Drug: Trametinib

INTERVENTIONS:
Drug: AMG 232 — Given an an oral tablet in escalating doses.
  Arms: AMG 232
Drug: Trametinib — Trametinib is an oral tablet given in a fixed dose.

SUMMARY:
Open-label, sequential dose escalation and expansion study of AMG 232 in subjects with acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years old
* Pathologically-documented, definitively-diagnosed AML that is relapsed or refractory to standard treatment, for which no standard therapy is available or the subject refuses standard therapy
* Ability to take oral medications and willing to record daily adherance to investigational product
* Adequate hematological, renal, hepatic, and coagulation laboratory assessments

Exclusion Criteria:

* Active infection requiring intravenous (IV) antibiotics
* Prior participation in an investigational study (procedure or device) within 21 days of study day 1
* Major surgery within 28 days of study day 1
* Anti-tumor therapy within 14 days of study day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of AMG 232 | 36 months
  To evaluate the safety and tolerability of AMG 232 by reviewing clinically significant or ≥ Grade 3 changes in safety laboratory tests, physical examinations, ECGs, or vitals signs in all subjects enrolled.
Characterize the pharmacokinetics of AMG 232 alone and in combination with trametinib when administered orally. | 36 months
  PK parameters will include, but are not limited to, area under the plasma concentration versus time curve (AUC) and Peak Plasma Concentration (Cmax).
Determine the maximum tolerated dose of AMG 232 alone and in combination with trametinib, if possible. | 36 months
  The MTD is defined at the highest dose level with an observed incidence of dose limiting toxicity in < 33% of subjects enrolled in a cohort.

SECONDARY OUTCOMES:
Treatment Response | 36 months
  Complete response (CR), complete response with incomplete recovery (CRi), and duration response.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Research Site, Birmingham, Alabama
  - Research Site, Buffalo, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington

REFERENCES:
- [Derived] Erba HP, Becker PS, Shami PJ, Grunwald MR, Flesher DL, Zhu M, Rasmussen E, Henary HA, Anderson AA, Wang ES. Phase 1b study of the MDM2 inhibitor AMG 232 with or without trametinib in relapsed/refractory acute myeloid leukemia. Blood Adv. 2019 Jul 9;3(13):1939-1949. doi: 10.1182/bloodadvances.2019030916. PMID 31253596
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com